CLINICAL TRIAL: NCT04035343
Title: Difference In Anatomic Integrity in Vitrectomy for Macula Off Rhegmatogenous RetiNal Detachments With Face Down Compared to Supine Positioning (the DIAMOND Study)
Brief Title: Effect of Type of Head Positioning on Retinal Displacement in Vitrectomy for Retinal Detachment
Acronym: DIAMOND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18-374
Record Dates: First submitted 2019-02-11; First posted 2019-07-29 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Retinal Detachment; Metamorphopsia
MeSH Terms: conditions — Retinal Detachment; Vision Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional face down positioning (Active Comparator): Patients in third arm will be treated with the current standard of care, that is, they will be kept supine in the ophthalmic surgery chair after the completion of their surgery. They will then be taken to the recovery area where, once transferred to the care of the postoperative care unit staff, they will transition to face down positioning. They will maintain this positioning until their first day postoperative visit after which they will position according to the retinal breaks found during surgery.
  Interventions: Behavioral: Face down positioning
- Supine positioning (Experimental): Patients in the second arm will be kept supine after the completion of their surgery. They will then be taken to the recovery area where, once transferred to the care of the postoperative care unit staff, they will maintain supine positioning. They will maintain this positioning until their first day postoperative visit after which they will position according to the retinal breaks found during surgery.
  Interventions: Behavioral: Supine positioning

INTERVENTIONS:
Behavioral: Face down positioning — See description of the face down positioning group
  Arms: Conventional face down positioning
Behavioral: Supine positioning — See description of the supine positioning group
  Arms: Supine positioning

SUMMARY:
Patients may experience metamorphopsia, or image distortion, after having vitrectomy to repair their rhegmatogenous retinal detachments especially those with a detached macula. Retinal displacement, as measured on autofluorescence photography, likely contributes to this distortion. It is thought that the retina slips inferiorly due to the residual subretinal fluid shifting as the patient transitions from the supine position intraoperatively to the sitting up position in the immediate postoperative period. By having the patient immediate position facedown or according to the retinal break, the risk of slippage is theoretically decreased.

DETAILED DESCRIPTION:
Rhegmatogenous retinal detachments (RRD) are a sight-threatening condition with an incidence of approximately 10 per 100 000 people. RRDs can be broadly classified into those with the macula still attached, and those with the macula detached. Visual prognosis for RRDs with attached macula tend to be much better than those with detached macula. Pars plana vitrectomy (PPV) is one of the procedures used to treat RRD. PPV is carried out in the operating room under regional anesthestic, and often times sedation. The retina is reattached by either draining the subretinal fluid through a peripheral retinal break, by draining the subretinal fluid through a posterior retinotomy, or by using a heavier-than-water liquid such as perfluorocarbon to push out the subretinal fluid. At the end of the surgery, the vitreous cavity is filled with a substance that will tamponade the retina to the wall of the eye. Tamponade agents can be temporary, such as sulfur hexafluoride (SF6) and octafluoropropane (C3F8), or long term, such as silicone oil. After the surgery, patients are usually told to put their facedown allowing the tamponade agent to keep the macula attached while the remaining subretinal fluid is reabsorbed by the retinal pigment epithelium. Alternatively, some surgeons ask that their patients position according to the location of their retinal breaks with the aim for the buoyant gas bubble to cover the break or breaks. Patients may experience metamorphopsia, or image distortion, after having their RRD repaired especially those with a detached macula. Retinal displacement, as measured on autofluorescence photography, likely contributes to this distortion. Supine positioning in theory covers all break locations as usually breaks occur in the anterior part of the retina near the vitreous base. This position has the advantage of being more ergonomic than face down. Depending on the results, this study might provide evidence for the current standard of care, which is face down positioning for the first day after vitrectomy for retinal detachment. Or, if supine positioning demonstrates superiority in reducing the risk of retinal displacement, patients would be able to maintain a more comfortable position after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Diagnosis of primary rhegmatogenous retinal detachment needing pars plana vitrectomy with the detachment involving at least one of the temporal vascular arcades, which would allow retinal displacement to be detected on fundus autofluorescence photography

Exclusion Criteria:

* Rhegmatogenous retinal detachment with an attached macula
* Proliferative retinopathy grade C or worst
* Prior vitrectomy for retinal detachment. Patients having had pneumatic retinopexy that failed to completely reattach the retina and therefore now needing vitrectomy are allowed into the study
* History of preoperative binocular diplopia
* Tamponade with silicone oil instead of gas
* Inability to maintain post operation head positioning
* Mental incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2019-08-26 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Retinal displacement | 3 months
  The presence of retinal vessels printing on fundus autofluorescence imaging.

SECONDARY OUTCOMES:
Visual Distortion | 3 months
  measured with M chart.
Aniseikonia | 3 months
  Measured with aniseikonia testing. The aniseikonia test measures the ratio of image size difference between the 2 eyes
Optical coherence tomography (OCT) changes | 3 months
  Changes seen on OCT
Optical coherence tomography angiography (OCTA) changes | 3 months
  Changes seen on OCTA
Metamorphopsia | 3 months
  Metamorphopsia is the image distortion experienced by the patient. It will be recorded in a data collection sheet as "yes" or "no" according to the patient subjective complain on metamorphopsia.
Best corrected Visual Acuity measured in "Early Treatment of Diabetic Retinopathy Study" letters | 3 months
  Best corrected Visual Acuity measured in "Early Treatment of Diabetic Retinopathy Study" letters

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, St. Michael's Hospital, Toronto, Ontario, Canada